CLINICAL TRIAL: NCT00327769
Title: A Double Blind, Double Dummy, Randomised, Multicentre Study to Compare the Efficacy and Safety of Fulvestrant 250mg With Arimidex 1mg as a Secondary-line Therapy in the Postmenopausal Women With Oestrogen Receptor Positive Advanced Breast Cancer
Brief Title: Faslodex Advanced Breast Cancer Local Chinese Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6997L00004
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced breast cancer; fulvestrant; anastrozole
MeSH Terms: interventions — Fulvestrant; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Anastrozole
  Interventions: Drug: Anastrozole
- 2 (Experimental): Anastrozole + Fulvestrant
  Interventions: Drug: Fulvestrant; Drug: Anastrozole

INTERVENTIONS:
Drug: Fulvestrant — 250 mg intramuscular injection
  Other Names: Faslodex; ZD9238
  Arms: 2
Drug: Anastrozole — 1 mg tablet
  Other Names: Arimidex; ZD1033

SUMMARY:
This study will evaluate the efficacy and safety of Faslodex as secondary-line treatment compared with Arimidex in oestrogen receptor positive postmenopausal advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal advanced breast cancer with oestrogen receptor positive
* Progression under first-line anti-oestrogen therapy.

Exclusion Criteria:

* Life-threatening metastasis; contraindication to anastrozole
* >2 regimens of hormonotherapy for advanced breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2005-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Time to Disease Progression (TTP)

SECONDARY OUTCOMES:
Objective Response Rate (ORR)
Clinical Benefit Rate (CBR)
Time to Treatment Failure (TTF)
Safety & Tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Breast Cancer Established Brands Team Medical Science Director, MD, Study Director — AstraZeneca
Locations (12):
- China (12):
  - Research Site, Beijing
  - Research Site, Dalian
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hankou
  - Research Site, Hefei
  - Research Site, Huangzhou
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Wuhan
  - Research Site, Xi'an

REFERENCES:
- [Derived] Xu B, Jiang Z, Shao Z, Wang J, Feng J, Song S, Chen Z, Gu K, Yu S, Zhang Y, Wang C, Zhang F, Yang J. Fulvestrant 250 mg versus anastrozole for Chinese patients with advanced breast cancer: results of a multicentre, double-blind, randomised phase III trial. Cancer Chemother Pharmacol. 2011 Jan;67(1):223-30. doi: 10.1007/s00280-010-1483-x. Epub 2010 Oct 12. PMID 20938664